CLINICAL TRIAL: NCT00087009
Title: Phase I Study of Oral ß-Glucan and Intravenous Rituximab Among Children and Adolescents With Relapsed CD20-Positive Lymphoma or Leukemia, or Post-Transplant Lymphoproliferative Disease
Brief Title: Beta-Glucan and Rituximab in Treating Young Patients With Relapsed or Progressive Lymphoma or Leukemia, or Lymphoproliferative Disorder Related to Donor Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-095; P30CA008748 (NIH); MSKCC-03095
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Leukemia; Lymphoma; Lymphoproliferative Disorder
Keywords: post-transplant lymphoproliferative disorder; recurrent childhood acute lymphoblastic leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence | interventions — beta-Glucans; Rituximab

ARMS (2):
- Group I (Experimental): Patients receive rituximab IV on days 1, 8, 15, and 22 and oral beta-glucan once daily on days 1-28 (days 8-28 of course 1). Treatment repeats every 42 days for 4 courses.
  Interventions: Biological: beta-glucan; Biological: rituximab
- Group II (Experimental): Patients receive rituximab IV on days 1, 4, 8, 15, and 22 and oral beta-glucan once daily on days 8-28. Beginning on day 42, patients with responding disease may receive monthly rituximab prophylaxis.
  Interventions: Biological: beta-glucan; Biological: rituximab

INTERVENTIONS:
Biological: beta-glucan — Given orally
Biological: rituximab — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Beta-glucan may increase the effectiveness of rituximab by making cancer cells more sensitive to the monoclonal antibody.

PURPOSE: This phase I trial is studying the side effects and best dose of beta-glucan when given together with rituximab in treating young patients with relapsed or progressive lymphoma or leukemia or with lymphoproliferative disorder related to donor stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of beta-glucan when given in combination with rituximab in pediatric patients with relapsed or progressive CD20-positive lymphoma or leukemia or post-allogeneic stem cell transplant-related lymphoproliferative disorder.
* Determine the toxicity of this regimen, with special emphasis on the degree of B-cell depletion and immune suppression, in these patients.
* Determine the effects of beta-glucan on leukocyte-mediated cytotoxic effects in patients treated with this regimen.

Secondary

* Determine the antitumor effect of this regimen in these patients.

OUTLINE: This is a dose-escalation study of beta-glucan. Patients are assigned to 1 of 2 treatment groups according to diagnosis.

* Group I (lymphoma or leukemia): Patients receive rituximab IV on days 1, 8, 15, and 22 and oral beta-glucan once daily on days 1-28 (days 8-28 of course 1). Treatment repeats every 42 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Group II (post-allogeneic stem cell transplant-related lymphoproliferative disorder): Patients receive rituximab IV on days 1, 4, 8, 15, and 22 and oral beta-glucan once daily on days 8-28. Beginning on day 42, patients with responding disease may receive monthly rituximab prophylaxis until their CD4 cell count is > 200/mm^3.

Cohorts of 6 patients receive escalating doses of beta-glucan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 6-24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * B-cell non-Hodgkin's lymphoma (NHL)
  * Hodgkin's lymphoma
  * Post-transplant lymphoproliferative disorder (PTLD)
  * Lymphoblastic leukemia
* CD20-positive disease verified by immunophenotyping at original diagnosis, disease relapse, or disease progression
* Refractory to conventional therapy, defined as 1 of the following:

  * Medically refractory HIV-associated NHL
  * Refractory or recurrent lymphoblastic leukemia
  * PTLD
  * In > first relapse or progression of B-cell NHL or Hodgkin's lymphoma
* Measurable (CT scan or MRI) or evaluable (marrow metastases or circulating lymphoblasts) disease within 4 weeks after completion of prior systemic (including systemic steroids) therapy

PATIENT CHARACTERISTICS:

Age

* Under 22

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 500/mm^3*
* Platelet count > 10,000/mm^3* NOTE: *Excluding patients with PTLD or CD20-positive lymphoblastic leukemia

Hepatic

* Hepatic toxicity ≤ grade 2

Renal

* Creatinine clearance ≥ 60 mL/min
* Renal toxicity ≤ grade 2

Cardiovascular

* Cardiac toxicity ≤ grade 2

Pulmonary

* Pulmonary toxicity ≤ grade 2

Immunologic

* Human anti-mouse antibody (HAMA) ≤ 1,000 units/mL
* Human anti-chimeric antibody titer negative
* No active, life-threatening infections except Epstein-Barr virus-associated lymphoproliferative disorder
* No history of allergy to mouse proteins
* No history of allergy to rituximab or other chimeric monoclonal antibodies
* No history of allergy to beta-glucan or oats, barley, mushrooms, or yeast

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Grade 3 hearing deficit allowed
* Gastrointestinal toxicity ≤ grade 2
* Neurologic toxicity ≤ grade 2
* No severe major organ toxicity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 4 weeks since prior rituximab
* No prior mouse antibodies
* No prior chimeric antibodies

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2004-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 2 years

SECONDARY OUTCOMES:
safety | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Nai-Kong V. Cheung, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Trudy N. Small, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States